CLINICAL TRIAL: NCT03060148
Title: The Treatment of Spinal Cord Stimulation in Severe Heart Failure
Brief Title: Spinal Cord Stimulation in Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMRPG3G0011
Record Dates: First submitted 2017-02-17; First posted 2017-02-23 (Actual); Last update posted 2017-06-09 (Actual); Status verified 2017-03

CONDITIONS: Heart Failure
Keywords: Heart failure; Spinal cord stimulation
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Medtronic neurostimulation
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Spinal cord stimulation (Active Comparator): Medtronic neurostimulation system for spinal cord stimulation
  Interventions: Device: Medtronic neurostimulation system
- Control (No Intervention): No implantation of Medtronic neurostimulation system

INTERVENTIONS:
Device: Medtronic neurostimulation system — Dual leads for spinal cord stimulation will be performed at 90% of the motor threshold for 24 hours/day at 50 Hz and pulse width 0.2 ms
  Other Names: Medtronic Restore Sensor™ Neurostimulation System
  Arms: Spinal cord stimulation

SUMMARY:
Previous studies have shown that spinal cord stimulation (SCS) may improve cardiac output and decrease the risk of ischemic ventricular arrhythmia in animal model and its safety profile in human trial. The purposes of this study are to evaluate the feasibility, treatment efficacy and safety of SCS in patients with severe symptomatic heart failure (HF).

DETAILED DESCRIPTION:
Morbidity and mortality in heart failure (HF) patients remain high, even with recent advances in therapies. Previous studies have shown that the autonomic nervous system plays an important role in the pathophysiology of HF and sudden cardiac death.

Spinal cord stimulation (SCS) is a neurostimulation therapy, which involves the stimulation of selected nerve fibers and intends to create end-organ responses characterized by changes in blood flow, decrease of catecholamines and reduction in inflammation. The SCS system consists of an implantable pulse generator (IPG) and dual leads. Each lead has electrodes on the distal end. Electrical impulses travel from the IPG through the leads to the electrodes positioned at the selected nerve fibers to provide the therapeutic stimulation. By virtue of its potential in augmenting blood flow, decreasing catecholamines and reducing inflammation, SCS may benefit HF patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients has a left ventricular ejection fraction between 20% and 35%
* Patient is in New York Heart Association Class III or in Ambulatory Class IV
* Patient is receiving stable medical therapy for HF (>90 days) at baseline
* Patient has a left ventricular end diastolic diameter between 55 mm and 80 mm
* Patient must be able and willing to provide written informed consent to participate in this study
* Patient must be able and willing to comply with the required follow-up schedule

Exclusion Criteria:

* Patient currently has an implanted spinal cord stimulator or previously had an implanted upper thoracic spinal cord stimulator which is now explanted
* Patient has polyneuropathy
* Patient requires short-wave diathermy, microwave diathermy or therapeutic ultrasound diathermy
* Patient has received a tissue/organ transplant (or is expected to have a tissue/organ transplant within the next 180 days)
* Patient has persistent or permanent atrial fibrillation
* Patient has chronic refractory angina or peripheral vascular pain
* Patient has critical valvular heart disease that requires valve repair or replacement
* Patient has had a myocardial infarction (MI) or cardiac revascularization procedure (percutaneous coronary intervention or coronary artery bypass graft) <90 days at baseline or is expected to have this in the next 180 days
* Patient is on IV inotropic therapy
* Patient has active myocarditis or early postpartum cardiomyopathy
* Patient has taken any of the following drugs within 30 days of enrollment: systemic corticosteroids, cytostatic and immunosuppressive drug therapy (cyclophosphamide, methotrexate, cyclosporine, azathioprine, etc.), DNA depleting or cytotoxic drugs
* Patient is pregnant, or of childbearing potential and is not using adequate contraceptive methods, or nursing
* Patient with a bleeding tendency (International Normalized Ratio >1.2 and platelet count <100 x10^9 per liter)
* Patient has a local infection at the implantable cardioverter-defibrillator (ICD) implant location or systemic infection
* Patient has renal insufficiency (creatinine >3.0 mg/dl)
* Patient is participating in another clinical study
* Patient is less than 20 years old
* Patient's life's expectancy is less than 1 years as assessed by investigator

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2017-06 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Composite of efficacy markers | 6 months
  Efficacy markers include peak oxygen uptake, New York Heart Association functional class, left ventricular structure and function (left ventricular end-systolic volume and ejection fraction), B-type natriuretic peptide, Minnesota Living with Heart Failure Questionnaire score: Improvement: +1; no change:0; worsening: -1.

SECONDARY OUTCOMES:
Post procedural adverse events | 24 months
  Post-procedure adverse events include implanted procedure related events, system related events and system modification related events.

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Li Wang, MD, Principal Investigator — Chang Gung Memorial Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zipes DP, Neuzil P, Theres H, Caraway D, Mann DL, Mannheimer C, Van Buren P, Linde C, Linderoth B, Kueffer F, Sarazin SA, DeJongste MJL; DEFEAT-HF Trial Investigators. Determining the Feasibility of Spinal Cord Neuromodulation for the Treatment of Chronic Systolic Heart Failure: The DEFEAT-HF Study. JACC Heart Fail. 2016 Feb;4(2):129-136. doi: 10.1016/j.jchf.2015.10.006. Epub 2015 Dec 9. PMID 26682789
- [Background] Tse HF, Turner S, Sanders P, Okuyama Y, Fujiu K, Cheung CW, Russo M, Green MDS, Yiu KH, Chen P, Shuto C, Lau EOY, Siu CW. Thoracic Spinal Cord Stimulation for Heart Failure as a Restorative Treatment (SCS HEART study): first-in-man experience. Heart Rhythm. 2015 Mar;12(3):588-595. doi: 10.1016/j.hrthm.2014.12.014. Epub 2014 Dec 12. PMID 25500165
- [Background] Lopshire JC, Zhou X, Dusa C, Ueyama T, Rosenberger J, Courtney N, Ujhelyi M, Mullen T, Das M, Zipes DP. Spinal cord stimulation improves ventricular function and reduces ventricular arrhythmias in a canine postinfarction heart failure model. Circulation. 2009 Jul 28;120(4):286-94. doi: 10.1161/CIRCULATIONAHA.108.812412. Epub 2009 Jul 13. PMID 19597055
- [Background] Foreman RD, Linderoth B, Ardell JL, Barron KW, Chandler MJ, Hull SS Jr, TerHorst GJ, DeJongste MJ, Armour JA. Modulation of intrinsic cardiac neurons by spinal cord stimulation: implications for its therapeutic use in angina pectoris. Cardiovasc Res. 2000 Aug;47(2):367-75. doi: 10.1016/s0008-6363(00)00095-x. PMID 10946073